CLINICAL TRIAL: NCT05481684
Title: The Importance of Embryo Transfer Day Progesterone Value in Natural Cycle Frozen Embryo Transfers and the Evaluation of the Effect of Rescue Therapy on Pregnancy Outcomes in Patients With Low Progesterone Levels: A Multicentric Randomized Controlled Study.
Brief Title: The Importance of Embryo Transfer Day Progesterone Value in Natural Cycle Frozen Embryo Transfers and the Evaluation of the Effect of Rescue Therapy on Pregnancy Outcomes in Patients With Low Progesterone Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26.07.2022-E.71262
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Infertility; IVF; Progesterone
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Progesterone group (Experimental): Progesterone level ≥ 10 ng/mL on ET day.
  Interventions: Other: Normal Progesterone group
- Low Progesterone group (Active Comparator): Progesterone level <10 ng/mL on ET day. Grup a Rescue vaginal progesterone, Grup b Rescue subcutan progesterone
  Interventions: Other: Low Progesterone group

INTERVENTIONS:
Other: Normal Progesterone group — No progesterone supplementation
  Arms: Normal Progesterone group
Other: Low Progesterone group — Progesterone level <10 ng/mL on ET day. If serum progesterone levels were <10 ng/ml at ET day, vaginal pills (Lutinus 2*1) or SC progesterone daily (Prolutex) was given to patients and ET was performed on the same day. Progesterone supplementation was discontinued if there was no pregnancy. Progesterone supplementation at the same dose was continued until 10 gestational weeks for viable pregnancies.
  Arms: Low Progesterone group

SUMMARY:
Thanks to recent advances in clinical practice and laboratory, embryo cryopreservation has become the first-line procedure in assisted reproductive technology. Improved laboratory techniques have increased the number of available embryos derived from an in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) cycle. Implementation of a single embryo transfer policy to improve vitrification, improve postwarm embryo survival rates, and reduce multiple pregnancies without reducing cumulative birth rates has contributed to an increase in the number of frozen-warms (1,2) Embryo freezing; It is becoming an adopted practice for an increasing number of indications, including prevention of ovarian hyperstimulation syndrome, preimplantation genetic testing (PGT), late follicular phase progesterone elevation, and embryo-endometrial asynchrony. In our study, we are investigating the effect of pre-transfer serum progesterone levels on pregnancy outcomes in patients who underwent frozen-thawed embryo transfer.Supplementary progesterone preparations can be used to prevent luteal phase defect and to provide progesterone support in cycle preparations for frozen-thawed embryo transfer(3). The aim in this study is to show the effect of serum progesterone level on the pregnancy results on the day of embryo transfer in natural cycles.

DETAILED DESCRIPTION:
The patients to be included in the study are the patients followed in the IVF centers of two different hospitals.Patients between the ages of 20-42 and having a BMI of <30, who are scheduled for IVF due to tubal factor, infertility of unknown cause, mild male factor, and anovulation will be included in the study. An antagonist (Cetrotide; Serono, Geneva, Switzerland) protocol will be used for controlled ovarian hyperstimulation, and recombinant follicle-stimulating hormone (recFSH) (Gonal F; Serono, Geneva, Switzerland) and Human Menopausal Gonadotropin (HMG) (Merional; Switzerland) will be used for stimulation. The dose of gonadotropin to be administered to patients is in the range of 150 to 450 IU per day and will be determined according to the age of each patient, serum FSH and E2 levels in the early follicular phase, and the number of antral follicles determined by ultrasound in the early follicular phase. Adjustment of the gonadotropin dose during the treatment will be adjusted by serial ultrasound measurements of the follicle diameters developed during the treatment and serum E2 levels. The patient's eggs will be collected at 34-36 hours. Fertilization check will be done the next day. During 3-5 days of embryo culture, embryo quality will be determined according to the D.Gardner criteria (1999). Embryos will be frozen on the 3rd or 5th day and transferred to a planned frozen cycle within the next month. In the frozen cycle, basal ultrasonography is performed on the 3rd day of the menstrual cycle and if there is no follicle over 10 mm, the patient will be called for a control on the 10th day of the cycle if the endometrial thickness is less than 5 mm. In the follow-ups after the 10th day, daily LH monitoring will be performed with the dominant follicle reaching 15 m in diameter. When the LH level increases 1.8 times, it will be considered as LH surge. Serum progesterone level will be checked on embrio transfer day. The patients with serum progesterone value below 10 on the day of embryo transfer will be divided into two groups, and the first group will be given vaginal progesterone (Lutinus 2*1) as rescue therapy, and the second group will be given subcutaneous progesterone (prolutex 1*1) as rescue therapy. Rescue treatment will not be applied to those whose serum progesterone level is 10 and above on the ET day. At the time of presumed LH surge, E2 (estradiol), P4 (progesterone), LH will be checked and the endometrial thickness in the uterus will be measured.

If the patient's endometrium is suitable, embryo transfer will be performed and a blood pregnancy test will be performed 10-12 days later. The research is planned to last for a year, starting in August 2022 and ending in August 2023. Patient data will be evaluated as prospective data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 20-42 who applied to the infertility clinic
* BMI<30

Exclusion Criteria:

* Severe male factor (Sperm count <5 ml/ml, progressively motile sperm count <10%)
* Intrauterine structural anomalies not corrected by surgery
* Hydrosalpenx if not underwent surgery
* Refusal to participate in the study
* cycle cancelation

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rates | average of 1 year
  fetal heartbeat by transvaginal ultrasound

SECONDARY OUTCOMES:
Ongoing pregnancy rate | average of 15 month
  Pregnancies that continue until the 12th week of pregnancy
Miscarriage | average of 15 month
  any clinical pregnancy lost before pregnancy week 12

CONTACTS AND LOCATIONS:
Overall Officials: pınar özcan, PhD, Principal Investigator — Bezmialem Foundation University; Cem Demirel, PhD, Study Chair — Acıbadem Ataşehir Hospital; Mehmet Erdem, PhD, Study Chair — Novaart IVF and Women's Health Center
Locations (3):
- Turkey (Türkiye) (3):
  - Acıbadem Ataşehir Hospital, Istanbul
  - Bezmialem Foundation University, Istanbul
  - Novaart IVF and Women's Health Center, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rienzi L, Gracia C, Maggiulli R, LaBarbera AR, Kaser DJ, Ubaldi FM, Vanderpoel S, Racowsky C. Oocyte, embryo and blastocyst cryopreservation in ART: systematic review and meta-analysis comparing slow-freezing versus vitrification to produce evidence for the development of global guidance. Hum Reprod Update. 2017 Mar 1;23(2):139-155. doi: 10.1093/humupd/dmw038. PMID 27827818
- [Result] Loutradi KE, Kolibianakis EM, Venetis CA, Papanikolaou EG, Pados G, Bontis I, Tarlatzis BC. Cryopreservation of human embryos by vitrification or slow freezing: a systematic review and meta-analysis. Fertil Steril. 2008 Jul;90(1):186-93. doi: 10.1016/j.fertnstert.2007.06.010. Epub 2007 Nov 5. PMID 17980870
- [Result] Groenewoud ER, Cohlen BJ, Macklon NS. Programming the endometrium for deferred transfer of cryopreserved embryos: hormone replacement versus modified natural cycles. Fertil Steril. 2018 May;109(5):768-774. doi: 10.1016/j.fertnstert.2018.02.135. PMID 29778369